CLINICAL TRIAL: NCT05387239
Title: Safety and Effectiveness of VL-PX10 + VL-P22 Treatment on Pulmonary Fibrosis Secondary to Covid-19
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor request
Sponsor: Vitti Labs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EW-02
Record Dates: First submitted 2022-05-16; First posted 2022-05-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pulmonary Fibrosis; COVID-19 Respiratory Infection
MeSH Terms: conditions — Pulmonary Fibrosis | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental/treatment arm (Experimental)
  Interventions: Drug: VL-PX10 and VL-P22 plus standard care
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VL-PX10 and VL-P22 plus standard care — The treatment consists of administration of VL-P22 and VL-PX10 plus standard care
  Arms: Experimental/treatment arm
Drug: Placebo — Saline plus standard care
  Arms: Placebo

SUMMARY:
The COVID-induced fibrotic lung damage continues long after viral infection has subsided and is exhibited by severe respiratory pathology and concomitant symptoms. The long-lasting sequelae in patients who have recovered from severe COVID indicate that there is a 30% chance of developing a persistent respiratory system pathology and a 10% chance of developing a severe pathology. The symptoms of lung fibrosis include a severe disruption of respiration, reduction of exercise tolerance, and concomitant development of persistent fibrotic lung damage. This study intends to evaluate benefits of a combination of VL-P22 and VL-PX10 in Covid-19 patients exhibiting pulmonary fibrosis.

DETAILED DESCRIPTION:
Multiple clinical trials are underway to explore options for treatment of pulmonary fibrosis in patients with history of COVID. Mesenchymal stem cell (MSC)-based therapies have been used worldwide for various pulmonary diseases. A recent review of over 110 reports of clinical trials worldwide with MSC-based therapies in pulmonary diseases found that these therapies have been reported to be safe and effective in the treatment of acute/viral pulmonary disease, community-acquired pneumonia (CAP), chronic obstructive pulmonary disease (COPD), bronchopulmonary dysplasia (BPD), interstitial lung diseases (ILD), chronic pulmonary fibrosis, bronchiolitis obliterans syndrome (BOS) and lung cancer. A phase 2 clinical trial in 101 severe Covid-19 patients with lung damage using human umbilical cord derived MSCs found that the treatment exerted numerical improvement in whole lung lesion volume and the 6-minute walk test from baseline to day 28 compared with the placebo.

This proof of concept, double-blind, placebo-controlled trial will evaluate the safety and efficacy of intravenous infusion of VL-PX10 and VL-P22, versus placebo, for use in the treatment of Covid induced Pulmonary Fibrosis. This is an add-on treatment study; subjects will be allowed to take standard of care treatments available.

The study will have two arms (n=10 each):

1. Experimental/treatment arm: VL-PX10 and VL-P22 plus standard care
2. Placebo: Saline plus standard care

The study duration would be 5 days of treatment plus 12 weeks follow up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible for enrollment in the study only if they meet the following criteria:

  1. Male or female, aged between 25 years (including) to 90 years old
  2. Confirmed and documented COVID-19 infection history with confirmed diagnosis of Pulmonary Fibrosis
  3. Negative to current Covid-19 infection as tested by RT-PCR/rapid antigen tests
  4. Able to perform a 6-minute walk test
  5. Blood routine, liver and kidney functions test values are within controllable range

     1. Adequate hepatic function as evidenced by ALT and AST < 2X ULN and bilirubin < 1.5X ULN for the reference lab
     2. Adequate renal function as evidenced by a serum creatinine ≤ 1.5 X ULN for the reference laboratory OR a calculated creatinine clearance of ≥ 60 mL/min by the Cockcroft-Gault Equation
     3. Adequate hematopoietic function as evidenced by white blood cells ≥ 3x109 / L and platelets ≥ 100x109 / L
  6. If childbearing age: agree to practice effective birth control from screening until 12 weeks after the last study treatment.

Exclusion Criteria:

* Subjects will be ineligible for enrollment in the study if they meet any of the following criteria:

  1. Clinically relevant heart condition such as, but not limited to, uncontrolled heart failure, severe pulmonary hypertension, atrial fibrillation or significant congenital heart disease
  2. Severe asthma on chronic therapy with biologics or steroids
  3. Active smokers as defined as individuals who currently smokes at least one cigarette or equivalent product a day. (Ex-smokers who had regularly smoked but who had not smoked the previous month are eligible)
  4. Evidence of active malignancy, or prior history of active malignancy not in remission.
  5. Life expectancy of < 6 months
  6. Patient included in another ongoing interventional therapeutic trial.
  7. Pregnant or Lactating.
  8. Serious or life-threatening co-morbidities, that in the opinion of the investigators, may compromise the safety or compliance with the study guidelines and tracking.

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate incidences of Treatment-Emergent Adverse Events following following VL-PX10 and VL-P22 administration to patients exhibiting Covid induced Pulmonary Fibrosis. | 3 months
  Presence of adverse events in less than 10% of the study population, as a measure of safety
To evaluate the efficacy of VL-PX10 and VL-P22 administration in alleviating long term symptoms of Covid induced Pulmonary Fibrosis, compared to placebo. | 3 months
  Change in distance walked on the six-minute walk test (6MWT). The 6MWT is a validated endpoint commonly used in clinical trial research.

SECONDARY OUTCOMES:
Change in Pulse Oximetry During the 6MWT | 3 months
  Oxygen saturation (pulse oximetry) during the 6-minute walk test (6MWT)
Incidence of Re-Hospitalization | 3 months
  Incidence of hospitalization after initial discharge and initiating treatment
Quality of Life assessment as collected using the SF-36 | 3 months
  The SF-36 (v2) is a self-administered questionnaire containing 36 items that measures functional status, well-being, and overall evaluation of health in 8 domains.

CONTACTS AND LOCATIONS:
Locations (1):
- Kit Bartalos, Liberty, Missouri, United States